CLINICAL TRIAL: NCT00459862
Title: Phase II Study of GW786034 in Patients With Malignant Pleural Mesothelioma
Brief Title: Pazopanib in Treating Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00656; NCI-2009-00656 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000539269; N0623 (Other: North Central Cancer Treatment Group); N0623 (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2013-10

CONDITIONS: Advanced Malignant Mesothelioma; Localized Malignant Mesothelioma; Recurrent Malignant Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant

ARMS (1):
- Arm I (Experimental): Patients receive 800 mg oral pazopanib hydrochloride once daily on days 1-21. Treatment repeats every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: laboratory biomarker analysis; Drug: pazopanib hydrochloride

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative study
Drug: pazopanib hydrochloride — Given orally

SUMMARY:
This phase II trial is studying the side effects and how well pazopanib works in treating patients with malignant pleural mesothelioma. Pazopanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the effect of pazopanib hydrochloride on the proportion of patients with malignant pleural mesothelioma who are progression-free at 6 months based on the RECIST criteria.

II. Determine the clinical toxicities of this drug in this patient population.

SECONDARY OBJECTIVES:

I. Determine the objective tumor response status in these patients as measured by the RECIST criteria or the modified RECIST criteria.

II. Determine the response rate in patients treated with this drug. III. Determine the effect of this drug on overall survival and time to progression in these patients.

IV. Assess predictive markers of activity of this drug in these patients. V. Assess serologic markers of target inhibition by this drug in these patients.

VI. Determine the clinical toxicities of this drug in this patient population.

OUTLINE: This is a multicenter study.

Patients receive oral pazopanib hydrochloride once daily on days 1-21. Treatment repeats every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.

Blood is collected at baseline and prior to each course of therapy and analyzed for markers of angiogenesis.

After completion of study therapy, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant pleural mesothelioma:

  * Measurable disease
  * No progressive disease inside or outside of any prior radiation field
* No symptomatic, untreated, or uncontrolled CNS metastases

  * Patients with CNS metastases treated with whole brain radiation (WBRT) may be enrolled after completion of WBRT

    * Patients may begin study therapy as early as the next day after completion of WBRT
* ECOG performance status 0-2
* Life expectancy >= 12 weeks
* ANC >=1,500/mm^3
* Platelet count >= 100,000/mm^3
* WBC >= 3,000/mm^3
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* AST and ALT =< 2.5 times ULN
* Alkaline phosphatase =< 2.5 times ULN
* Creatinine =< 1.5 times ULN or creatinine clearance >= 50 mL/min
* Proteinuria =< 1+ on 2 consecutive dipsticks taken >= 1 week apart
* No condition that impairs ability to swallow and retain study drug tablets including, but not limited to, any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication
  * Requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* No other primary malignancy except for carcinoma in situ of the cervix or nonmelanomatous skin cancer, unless that prior malignancy was diagnosed and definitively treated ≥ 5 years ago with no subsequent evidence of recurrence
* Patients with a history of low-grade (Gleason score =< 6) localized prostate cancer are eligible even if diagnosed within the past 5 years
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to pazopanib hydrochloride or other agents used in the study
* None of the following concurrent severe and/or uncontrolled medical conditions:

  * Serious or nonhealing wound, ulcer, or bone fracture
  * Abdominal fistula, diverticulosis, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
  * Poorly controlled diabetes
  * Interstitial pneumonia
  * Extensive and symptomatic interstitial fibrosis of the lung
* No cardiovascular illness or complication, including any of the following:

  * Any history of cerebrovascular accident within the past 6 months
  * History of myocardial infarction (prior electrocardiographic evidence of myocardial injury)
  * History of cardiac arrhythmia (prior electrocardiographic evidence of abnormal heart rhythm)
  * Admission for unstable angina
  * Cardiac angioplasty or stenting within the past 12 months
  * NYHA class III-IV heart failure

    * Asymptomatic NYHA class II heart failure allowed
  * QTc prolongation (defined as a QTc interval ≥ 500 msecs) or other significant electrocardiogram abnormalities
  * Venous thrombosis within the past 12 weeks
* No ancillary therapy considered investigational within the past 4 weeks
* No symptomatic, untreated, or uncontrolled seizure disorder
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit study compliance
* No significant traumatic injury within the past 4 weeks
* No more than 1 prior systemic therapy for malignant pleural mesothelioma
* No major surgery (i.e., laparotomy) or open biopsy within the past 4 weeks

  * Insertion of a vascular access device is not considered major or minor surgery
* No minor surgery within the past 2 weeks

  * Insertion of a vascular access device is not considered major or minor surgery
* Prior palliative radiotherapy allowed

  * No prior palliative radiotherapy to the chest except for a maximum of 3 fractions of radiotherapy for superior vena cava syndrome
* No concurrent therapeutic warfarin

  * Low molecular-weight heparin or prophylactic low-dose warfarin allowed
* No other concurrent chemotherapy, immunotherapy, hormonal therapy, or radiotherapy
* No concurrent medications that act through the CYP450 system
* No concurrent combination antiretroviral therapy for HIV-positive patients
* PT/INR/PTT =< 1.2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception
* No uncontrolled infection
* No uncontrolled blood pressure (BP) (defined as systolic BP > 140 mm Hg and/or diastolic BP > 90 mm Hg in spite of adequate anti-hypertensive therapy)
* No other severe underlying disease that, in the judgment of the investigator, would limit study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-03; Primary Completion 2009-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Molina, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Parikh K, Mandrekar SJ, Allen-Ziegler K, Esplin B, Tan AD, Marchello B, Adjei AA, Molina JR. A Phase II Study of Pazopanib in Patients with Malignant Pleural Mesothelioma: NCCTG N0623 (Alliance). Oncologist. 2020 Jun;25(6):523-531. doi: 10.1634/theoncologist.2019-0574. Epub 2019 Dec 24. PMID 31872928

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-four participants were accrued between May 2007 and October 2008.
Pre-assignment Details: All 34 participants were evaluable for the primary endpoint.
Groups:
- Arm I: Patients receive 800mg oral pazopanib hydrochloride once daily on days 1-21. Treatment repeats every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients receive oral pazopanib hydrochloride once daily on days 1-21. Treatment repeats every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 73 [49 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Evaluable Participants Who Are Progression-free at 6 Months Based on the Response Evaluation Criteria for Solid Tumors (RECIST)
Description: The proportion of patients who are progression-free at 6 months is calculated by dividing the number of evaluable participants who are progression-free at 6 months based on the Response Evaluation Criteria for Solid Tumors (RECIST) by the total number of evaluable participants.
Time Frame: 6 months
Population: All 34 participants were analyzed for this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 34
percentage of participants | 47.8

2. Secondary Outcome: Overall Survival
Time Frame: From study enrollment to time of death from any cause or censored at last follow-up, up to 3 years
Population: All 34 participants were evaluable for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 34
months | 11.5 [6.2 to 18.2]

3. Secondary Outcome: Progression-free Survival Assessed by RECIST
Time Frame: From study enrollment to the first date of disease progression or death as a result of any cause, whichever occurs first, up to 3 years
Population: All 34 participants were analyzed for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 34
months | 4.2 [2.5 to 5.9]

4. Secondary Outcome: Determine the Clinical Toxicities of This Drug in This Participant Population.
Description: The number of participants with a reported Grade 3, Grade 4, and Grade 5 toxicity, regardless of attribution, will be tabulated.
Time Frame: Participants will be evaluated every cycle during treatment
Population: All 34 participants were evaluable for adverse events.
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 34
participants
  Grade 3 or Higher | 23
  Grade 4 or Higher | 5
  Grade 5 | 3

5. Secondary Outcome: Overall Best Response of Target Lesions to Pazopanib in Patients With MPM Based on the RECIST.
Description: Complete Response (CR): Disappearance of all target lesions.
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline LD.
Time Frame: From study enrollment to the first date of disease progression
Population: All 34 participants were evaluable for this endpoint.
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 34
participants
  Partial Response (PR) | 5
  Complete Response (CR) | 0

6. Secondary Outcome: Overall Response Rate
Description: To evaluate the confirmed response rate of pazopanib in patients with MPM based on the RECIST criteria for MPM. Responses are confirmed by repeat assessments that are be performed no less than 4 weeks after the criteria for response are first met.
  Complete Response (CR): Disappearance of all target lesions.
  Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: Participants will be evaluated every cycle during treatment, up to 2 years
Population: All 34 participants were evaluable for this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm I
Number analyzed (Participants) | 34
percentage of patients | 5.9 [0.7 to 19.7]

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 13/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=34)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Taste alteration (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=34)
Hemoglobin decreased (Blood and lymphatic system disorders) | 17 (69)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (6)
Vision blurred (Eye disorders) | 1 (4)
Watering eyes (Eye disorders) | 2 (7)
Abdominal pain (Gastrointestinal disorders) | 16 (42)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 15 (55)
Dry mouth (Gastrointestinal disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 3 (7)
Flatulence (Gastrointestinal disorders) | 2 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroscopy abnormal (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 19 (65)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 12 (23)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 27 (156)
Pneumonia (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 19 (44)
Alkaline phosphatase increased (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 19 (47)
Bilirubin increased (Investigations) | 5 (18)
Leukocyte count decreased (Investigations) | 11 (26)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 5 (6)
Platelet count decreased (Investigations) | 10 (23)
Weight loss (Investigations) | 3 (7)
Anorexia (Metabolism and nutrition disorders) | 13 (30)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (6)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 1 (2)
Memory impairment (Nervous system disorders) | 1 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (30)
Syncope (Nervous system disorders) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 10 (37)
Anxiety (Psychiatric disorders) | 4 (10)
Confusion (Psychiatric disorders) | 1 (4)
Depression (Psychiatric disorders) | 2 (4)
Insomnia (Psychiatric disorders) | 2 (3)
Proteinuria (Renal and urinary disorders) | 13 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (6)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (5)
Rash desquamating (Skin and subcutaneous tissue disorders) | 12 (32)
Hypertension (Vascular disorders) | 27 (70)
Vascular disorder (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less